CLINICAL TRIAL: NCT05496205
Title: A Randomized, Double-blind, Placebo-controlled, Single- Ascending Dose Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics/Pharmacodynamics Properties of iN1011-N17 After Oral Administration in Healthy Volunteers
Brief Title: A SAD Study to Evaluate the Safety, Tolerability and PK/PD of iN1011-N17 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: iN Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP17061101
Record Dates: First submitted 2022-05-30; First posted 2022-08-11 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis; Pain; Post Herpetic Neuralgia; Neuropathic Pain; Chronic Pain; Nav 1.7
Keywords: Nav1.7 Inhibitor; Neuropathic pain; Postoperative pain; Chemotherapy-induced neuropathic pain; Nav 1.7; Pain; Sodium Channel; Volatage Gated Sodium Channel; Voltage Gated Sodium Channel 1.7; DRG Voltage Gated Sodium Channel 1.7; Sodium Channel 1.7
MeSH Terms: conditions — Osteoarthritis; Pain; Neuralgia, Postherpetic; Neuralgia; Chronic Pain; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- iN1011-N17, Oral capsule, Single Ascending Dose (Experimental): The IP or placebo will be orally administered in the morning on Day 1, following a 10-hour overnight fast.
  Interventions: Drug: iN1011-N17
- iN1011-N17, Oral Suspension, Single Ascending Dose (Experimental): The IP or placebo will be orally administered in the morning on Day 1, following a 10-hour overnight fast.
  Interventions: Drug: iN1011-N17
- iN1011-N17, Nanoparticle Capsule, Single Ascending Dose (Experimental): The IP or placebo will be orally administered in the morning on Day 1, following a 10-hour overnight fast.
  Interventions: Drug: iN1011-N17
- Placebo (Placebo Comparator): The IP or placebo will be orally administered in the morning on Day 1, following a 10-hour overnight fast.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: iN1011-N17 — This study will be conducted in approximately 104 healthy subjects in up to 13 sequential dose cohorts. Thirteen cohorts will consist of up to 8 subjects, including 2 subjects receiving placebo and 6 subjects receiving iN1011-N17.
  Each subsequent cohort will continue to be randomized and dosed until maximum exposure is attained or a stopping criterion has been reached.
  Arms: iN1011-N17, Nanoparticle Capsule, Single Ascending Dose; iN1011-N17, Oral Suspension, Single Ascending Dose; iN1011-N17, Oral capsule, Single Ascending Dose
Drug: Placebo — Matching Placebo for each formulations
  Arms: Placebo

SUMMARY:
A First-in-Human, Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics/Pharmacodynamics of iN1011-N17 after Oral Administration in Healthy Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female adults aged 18 to 55 years (inclusive at the time of written informed consent).
2. Body mass index (BMI = body weight (kg)/[height (m)]2) between 18 kg/m2 and 32 kg/m2 (inclusive) at the time of Screening, and a minimum weight of 50 kg.
3. Clinical laboratory values within normal range as specified by the testing laboratory at Screening and Day -1, unless deemed not clinically significant by the Investigator.
4. Clinically acceptable blood pressure (BP), pulse, respiratory rate (RR), and body temperature (SBP between 90 and 140 mmHg; DBP between 40 and 90 mmHg; pulse between 40 and 100 bpm; RR between 10 and 22 breaths/min; body temperature between 35.5°C and 37.5°C) at Screening and Day -1. Measurements are to be recorded after a minimum of 5 minutes of resting in sitting or supine position.
5. Female subjects must be of non-child-bearing potential, defined as:

   1. Surgically sterile (i.e., had a bilateral tubal ligation, hysterectomy, salpingectomy, or bilateral oophorectomy at least 6 months before the first dose of investigational product [IP]) or;
   2. Postmenopausal for at least 1 year before the first dose of IP, and if they have follicle-stimulating hormone (FSH) levels in the postmenopausal range for the investigational site/institution.

   OR

   Female subjects of child-bearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Day -1, and must not be breastfeeding, lactating or planning pregnancy during the study period.

   Female subjects must agree to use adequate contraception from Screening until 30 days after the last dose of IP.

   Adequate contraception is defined as a condom for the male partner combined with either:
   1. Non-hormonal intrauterine device (IUD)
   2. Vasectomized partner with documented azoospermia 90 days after procedure, if that partner is the sole sexual partner

   Male subjects who are sexually active must use a condom combined with use of a highly-effective method of contraception for the female partner. Acceptable highly-effective forms of contraception for partners of male subjects are as follows:
   1. Hormonal methods of contraception including oral contraceptives containing estrogen and progesterone, a vaginal ring, injectable and implantable hormonal contraceptives, intrauterine hormone-releasing system (e.g. Mirena) and progesterone-only hormonal contraception associated with inhibition of ovulation.
   2. Non-hormonal intrauterine device (IUD).
   3. Bilateral tubal occlusion.
   4. Surgically sterile.
   5. Post-menopausal status. Male subjects must continue to use adequate contraception, as well as refrain from donating sperm for 90 days after the last dose of IP.

   Complete abstinence is an acceptable form of contraception where it is the usual and preferred lifestyle.

   Subjects who are exclusively in same-sex relationships are not required to use contraception, however, males should refrain from donating sperm for 90 days after the last dose of IP and females should refrain from donating ova or undergoing fertility treatment for 30 days following the last dose of IP.
6. Cognitively capable of understanding the provided information and able to fully comply with protocol requirements.
7. Written informed consent prior to the commencement of any study procedures.
8. Willing and able to perform the necessary visits to the investigational site/institution.
9. In good general health at the Investigator's discretion, with no significant medical history, and with no clinically significant abnormalities on physical examination at Screening and before the first dose of IP.

Exclusion Criteria:

1. Presence or history of hepatic, renal, neurological, pulmonary, endocrine, hematologic, cardiovascular or genitourinary disease that, in the opinion of the Investigator, may affect the evaluation of the investigational product or place the participant at undue risk.
2. Presence of any underlying physical or psychiatric condition that, in the opinion of the Investigator, would undermine subject compliance to protocol requirements.
3. Presence or history of gastrointestinal disease (e.g., peptic ulcer, gastritis, gastric cramp, gastroesophageal reflex disease, Crohn's disease) or history of gastrointestinal surgery (except simple appendectomy or herniorrhaphy) that may affect assessment of safety and pharmacokinetic characteristics of the IP.
4. History of hypersensitivity to iN1011-N17 or to any of its components.
5. History of allergy or sensitivity to sulfonamides.
6. Any abnormal 12-lead ECG findings at Screening and Day -1, deemed by the Investigator or designee to be clinically significant.
7. Positive test for HBsAg, HCV, or HIV at Screening.
8. Positive urine drug screen test (including: amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine, phencyclidine and tetrahydrocannabinol) or alcohol breath test at Screening and Day -1.
9. History of fracture or other significant injury to dominant arm or current injury or condition, such as carpel tunnel syndrome, that may prevent accurate sensory testing.
10. Use of any prescription drugs within 14 days and for OTC medications, herbal remedies (including St John's Wort), dietary supplements or vitamins within 7 days, or five half-lives of the product, whichever is longer, before the first dose of IP and for the duration of the study without prior approval of the Investigator and the MM. This includes analgesics such as paracetamol and non-steroidal anti-inflammatories.
11. The use of any IP or investigational medical device within 30 days prior to Screening, or five half-lives of the product, whichever is longer.
12. Blood or plasma donation of more than 450 mL within 90 days before the first dose of IP and for the duration of the study. It is recommended that blood/plasma donations not be made for at least 30 days after study completion.
13. History of alcoholism, substance or drug abuse-related disorders deemed significant by the Investigator (or designee) (i.e. >21 units per week for males and >14 units per week for females. One unit of alcohol equals ½ pint [285 mL] of beer or lager, 1 glass [125 mL] of wine, or 1/6 gill [25 mL] of spirits).
14. Use of more than five nicotine-based products (including smoking tobacco, smokeless tobacco, and nicotine patches) per week, within 90 days prior to Screening. Subjects must have a negative urine cotinine test at both Screening and Day -1 and refrain from the use of any nicotine-based products for the duration of the study.
15. Consumption of beverages or foods that contain grapefruit, star fruit, pomelos, or products containing these fruits, from 7 days, or from the time that is deemed significant by the investigator, and products containing caffeine (e.g., coffee, green tea, black tea and sodas) from 72 hours before the first dose of IP until discharge from the unit.
16. Unwilling to refrain from strenuous exercise from 48 hours prior to admission to the investigational site/institution and for the duration of the study, where strenuous exercise is defined as that which requires significant effort, energy, or strength, such as lifting weights or running.
17. Any other reason that, in the opinion of the Investigator, may affect assessment of safety, PK or PD characteristics of the IP.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and causality of adverse events (AEs) and serious adverse events (SAEs) | Day 1 to Day 8
Number of participants with abnormal physical examination findings | Screening, Day -1, Day 3, Day 8
  Full physical examination will consist of the following body systems: general appearance, HEENT (head, ears, eyes, nose, and throat), cardiovascular, respiratory system, abdomen, musculoskeletal, neurological, lymph nodes, skin, and other.
Vital Signs (Blood Pressure) | Screening, Day -1, Day 1 (pre-dose and 2, 4, 8 hours pose-dose), Day 2 (prior PK sampling), Day 3 (prior PK sampling), Day 8
  Vital signs (BP) will be listed and summarized at each protocol specified time point. Observed and change from baseline will be summarized at each protocol specified time point.
Vital Signs (Pulse) | Screening, Day -1, Day 1 (pre-dose and 2, 4, 8 hours pose-dose), Day 2 (prior PK sampling), Day 3 (prior PK sampling), Day 8
  Vital signs (Pulse) will be listed and summarized at each protocol specified time point. Observed and change from baseline will be summarized at each protocol specified time point.
Vital Signs (Respiratory Rate) | Screening, Day -1, Day 1 (pre-dose and 2, 4, 8 hours pose-dose), Day 2 (prior PK sampling), Day 3 (prior PK sampling), Day 8
  Vital signs (RR) will be listed and summarized at each protocol specified time point. Observed and change from baseline will be summarized at each protocol specified time point.
Vital Signs (Body temperature) | Screening, Day -1, Day 3 (prior PK sampling), Day 8
  Vital signs (Body temperature) will be listed and summarized at each protocol specified time point. Observed and change from baseline will be summarized at each protocol specified time point.
12-lead electrocardiogram(ECG) | Screening, Day -1, Day 1 (pre-dose and 1, 4, 8 hours pose-dose), Day 3 (prior PK sampling), Day 8
  ECG values will consist of QT interval, PR interval, QRS interval, RR interval and QTcF. Values will be listed and summarized at each protocol specified time point. Observed and change from baseline will be summarized at each protocol specified time point.
Number of participants with abnormal Laboratory tests (Hematology) | Screening, Day -1, Day 3 prior to discharge, Day 8
  Laboratory evaluations will be listed and summarized for each scheduled visit. Observed and change from baseline clinical laboratory data will be summarized at each protocol specified time point.
Number of participants with abnormal Laboratory tests (Biochemistry)) | Screening, Day -1, Day 3 prior to discharge, Day 8
  Laboratory evaluations will be listed and summarized for each scheduled visit. Observed and change from baseline clinical laboratory data will be summarized at each protocol specified time point.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 0-48 hours post dose
Time to maximum plasma concentration (tmax) | 0-48 hours post dose
Terminal half-life (t1/2) | 0-48 hours post dose
Area under the plasma concentration curve (AUClast, AUCinf) | 0-48 hours post dose
Apparent volume of distribution (Vz/F) | 0-48 hours post dose on Day 1 to Day 3
Apparent plasma elimination rate constant (λz) | 0-48 hours post dose on Day 1 to Day 3
Apparent clearance (CL/F) | 0-48 hours post dose on Day 1 to Day 3
Fraction excreted unchanged in urine (fe) | 0-48 hours post dose on Day 1 to Day 3
Amount of drug excreted unchanged in the urine (Ae) | 0-48 hours post dose on Day 1 to Day 3
Renal clearance (CLR) | 0-48 hours post dose on Day 1 to Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia